CLINICAL TRIAL: NCT03012308
Title: Evaluation of Left Ventricular Filling Pressures in Post-operative Cardiac Surgery: Trans-thoracic Ultrasound VS Invasive Pressure of the Left Atrium
Brief Title: Trans-thoracic Ultrasound VS Invasive Pressure of the Left Atrium
Acronym: ECHOPOG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6655 - ECHOPOG
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-01

CONDITIONS: Myocardial Dysfunction
Keywords: Myocardial Dysfunction; left ventricular; mitral valve doppler; mitral ring doppler; ultrasound signs; lung edema
MeSH Terms: conditions — Pulmonary Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As part of cardiac and hemodynamic evaluation of patients, echocardiographic measurements allow indirect evaluation of left ventricular filling pressures (LVFP). These ultrasound parameters, including mitral valve doppler and mitral ring doppler (in particular the E / E 'ratio), are well validated in medical cardiology and in some resuscitation patients. The measurement of filling pressures is an important daily element in the medical management of patients in intensive care, in particular on the hemodynamic and respiratory levels. No studies have evaluated the relevance of these markers in a postoperative context of cardiac surgery. Indeed, the surgery alters the cardiac function, which could modify the values of the echocardiographic parameters and their predictability. Left atrium pressure (LAP) directly reflects LVFP and is measured in cardiac surgical resuscitation by a surgically placed catheter as part of routine institutional care and will serve as gold-standard. To study the clinical significance of these LAP and LVFP values estimated by cardiac ultrasound, we will study their correlation with clinical and ultrasound signs of acute lung edema (ALE).

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in surgical resuscitation for cardiac surgery with heart-lung bypass machine

Exclusion Criteria:

* No consent
* Mitral valve surgery
* severe MI / severe mitral narrowing.
* Absence of POG catheter
* Urgent surgery
* Heart transplant / mechanical assistance
* Classics: minors, pregnant women, guardianship / curatorship / safeguarding,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient hospitalized in surgical resuscitation for cardiac surgery with heart-lung bypass machine, aged over 18 years
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-12-20 (Actual); Primary Completion 2017-12-20 (Estimated); Study Completion 2017-12-20 (Estimated)

PRIMARY OUTCOMES:
Compare the mean values of LAP between the group "high filling pressures" and the group "non-high filling pressures" | 6 postoperative hours of cardiac surgery of patients hospitalized in surgical resuscitation

CONTACTS AND LOCATIONS:
Overall Officials: Gharib AJOB, MD, Study Director — University Hospital, Strasbourg, France; Paul-Michel MERTES, MD, PhD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Service Réanimation chirurgicale cardio-vasculaire - NHC, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No